CLINICAL TRIAL: NCT01266967
Title: BRF113929: An Open-Label, Two-Cohort, Multicentre Study of GSK2118436 as a Single Agent in Treatment Naïve and Previously Treated Subjects With BRAF Mutation-Positive Metastatic Melanoma to the Brain
Brief Title: A Study of GSK2118436 in BRAF Mutant Metastatic Melanoma to the Brain
Acronym: Break MB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113929
Record Dates: First submitted 2010-12-02; First posted 2010-12-24 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-03

CONDITIONS: Melanoma and Brain Metastases
Keywords: GSK2118436; Metastatic melanoma to the brain; Brain metastases; Braf mutation; Brain neoplasm; BRAF inhibitor
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Single arm with 2 cohorts; Cohort A no previous brain therapy and Cohort B previous brain therapy
  Interventions: Drug: GSK2118436

INTERVENTIONS:
Drug: GSK2118436 — Subjects in this study receive 150 mg of GSK2118436 twice daily and continue on treatment until disease progression, death, or unacceptable adverse event.
  Other Names: Dabrafenib

SUMMARY:
This study is designed to assess the efficacy, pharmacokinetics, safety, and tolerability of an oral, twice daily dose of 150 mg GSK2118436 administered to subjects with BRAF V600E or V600K mutation-positive metastatic melanoma to the brain. Subjects in Cohort A will not have received any local brain therapy, and subjects in Cohort B will have received prior local therapy for brain metastases. Subjects will continue on treatment until disease progression, death, or unacceptable adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A:
* No prior local therapy for brain metastases.
* Subjects who are receiving concomitant corticosteroids must be on a stable or decreasing dose for at least 3 weeks prior to first dose of study treatment.
* No prophylactic or preventive anti-epileptic therapy. Exception: anti-epileptic therapy indicated in order to prevent neurologic symptoms caused by a pre-existing condition and not related to brain metastasis is allowed.
* Cohort B:
* Subjects must have received at least one local therapy for brain metastases including but not restricted to brain surgery, Whole Brain Radiotherapy or Stereotactic Radiosurgery (e.g. gamma knife, linear-accelerated-based radiosurgery, charged particles, and CyberKnife). Multiple local therapies or combinations of local therapies are allowed. For subjects receiving local therapy to all brain lesions (including WBRT), progression of pre-existing lesions based on RECIST 1.1 (> 20% increase in longest diameter on baseline scan) or new measurable lesions are required. For subjects receiving local therapy for some but not all lesions, disease progression based on RECIST 1.1 is not required as long as there are remaining brain lesions that are measurable and not previously treated.
* Subjects who are receiving concomitant corticosteroids must be on a stable or decreasing dose for at least 2 weeks prior to first dose of study treatment.
* Prophylactic or preventive anti-epileptic therapy is allowed.
* General:
* Must sign written informed consent.
* Must be at least 18 years of age.
* Histologically confirmed metastatic melanoma (Stage IV), carrying BRAF V600E- or V600K-mutation.
* Up to two previous treatment regimens for extracranial metastatic melanoma including chemo-, cytokine-, immuno-, biological- and vaccine-therapy.
* At least one measurable intracranial target lesion for which all of the following criteria have to be met:
* previously untreated or progressive according to RECIST 1.1 (greater than or equal to 20% increase in longest diameter on baseline scan) after previous local therapy
* immediate local therapy clinically not indicated or patient is not a suitable candidate to receive immediate local therapy
* largest diameter of greater than or equal to 0.5cm but less than or equal to 4 cm as determined by contrast-enhanced MRI
* for target lesions (for definition see Section 6.1.1) with diameter of greater than 0.5 cm but less than or equal to 1 cm documented measurement by a neuroradiologist is required.
* for all lesions with diameter of greater than or equal to 3 cm but less than or equal to 4 cm documented measurement by a neuroradiologist is required.
* Time interval between last day of previous anti-tumour systemic treatment and first dose of GSK2118436:
* 14 days elapsed from last treatment with surgery, SRS or gamma knife
* 28 days elapsed from last treatment with WBRT
* Greater than or equal to 28 days or five half-lives (whichever is longer) have elapsed from last dose of approved or investigational chemo-, cytokine-, immune-, biological-, or vaccine-therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Adequate organ function.
* Women with child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control during the study.
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to the first dose of study treatment.

Exclusion Criteria:

* Neurological symptoms related to brain metastasis.
* Previous treatment with a BRAF or MEK inhibitor.
* Current or expected use of a prohibited medication during treatment with GSK2118436.
* Presence of leptomeningeal disease or primary dural metastases.
* Known allergies against contrast agents required for magnetic resonance imaging (MRI) of intracranial lesions.
* Current use of therapeutic warfarin. NOTE: Low molecular weight heparin and prophylactic low-dose warfarin are permitted.
* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI v4.0) Grade 2 or higher from previous anti-cancer therapy, except alopecia.
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption of drugs.
* A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection.
* Acute infection requiring intravenous antibiotics
* History of another malignancy. Exception: (a) Subjects who have been disease-free for 5 years, (b) a history of completely resected non-melanoma skin cancer, (c) successfully treated in situ carcinoma, (d) CLL in stable remission, or (e) indolent prostate cancer requiring no or only anti-hormonal therapy with histologically confirmed tumour lesions that can be clearly differentiated from melanoma target and non-target lesions are eligible.
* Certain cardiac abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- United States (8):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Seattle, Washington
- Australia (3):
  - GSK Investigational Site, Waratah, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (4):
  - GSK Investigational Site, Boulogne-Billancourt
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Villejuif
- Germany (3):
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Italy (2):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Padua, Veneto

REFERENCES:
- [Background] Long GV, Trefzer U, Davies MA, Kefford RF, Ascierto PA, Chapman PB, Puzanov I, Hauschild A, Robert C, Algazi A, Mortier L, Tawbi H, Wilhelm T, Zimmer L, Switzky J, Swann S, Martin AM, Guckert M, Goodman V, Streit M, Kirkwood JM, Schadendorf D. Dabrafenib in patients with Val600Glu or Val600Lys BRAF-mutant melanoma metastatic to the brain (BREAK-MB): a multicentre, open-label, phase 2 trial. Lancet Oncol. 2012 Nov;13(11):1087-95. doi: 10.1016/S1470-2045(12)70431-X. Epub 2012 Oct 8. PMID 23051966
- [Derived] Santiago-Walker A, Gagnon R, Mazumdar J, Casey M, Long GV, Schadendorf D, Flaherty K, Kefford R, Hauschild A, Hwu P, Haney P, O'Hagan A, Carver J, Goodman V, Legos J, Martin AM. Correlation of BRAF Mutation Status in Circulating-Free DNA and Tumor and Association with Clinical Outcome across Four BRAFi and MEKi Clinical Trials. Clin Cancer Res. 2016 Feb 1;22(3):567-74. doi: 10.1158/1078-0432.CCR-15-0321. Epub 2015 Oct 7. PMID 26446943
- [Derived] Ouellet D, Gibiansky E, Leonowens C, O'Hagan A, Haney P, Switzky J, Goodman VL. Population pharmacokinetics of dabrafenib, a BRAF inhibitor: effect of dose, time, covariates, and relationship with its metabolites. J Clin Pharmacol. 2014 Jun;54(6):696-706. doi: 10.1002/jcph.263. Epub 2014 Jan 17. PMID 24408395

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK2118436 150 mg: No Prior Local Therapy: Participants who received no prior local therapy for brain metastasis received GSK2118436 150 milligram (mg) capsules either one hour before or 2 hours after a meal twice daily until evidence of disease progression, death, or unacceptable adverse events.
- GSK2118436 150 mg: Prior Local Therapy: Participants who received prior local therapy for brain metastasis received GSK2118436 150 mg capsules either one hour before or 2 hours after a meal twice daily until evidence of disease progression, death, or unacceptable adverse events.
Period: Overall Study
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Started | 89 | 83
Completed | 0 | 0
Not Completed | 89 | 83
Not completed — Death | 69 | 61
Not completed — Study Closed/Terminated | 15 | 17
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy | Total
Number analyzed (Participants) | 89 | 83 | 172
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (13.35) | 52.7 (13.83) | 52.5 (13.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 65 | 55 | 120
Race/Ethnicity, Customized [Number; unit: participants] — Race was not reported for one participant who recevied prior local therapy.
  participants
    White | 89 | 82 | 171
    Not reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With BRAF V600E Mutation-positive Melanoma With Overall Intracranial Response (OIR), as Assessed by the Investigator
Description: OIR is defined as the number of participants whose intracranial response was a confirmed complete response (CR) or partial response (PR) assessed by investigators using modified Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. CR is defined as disappearance of all lesions. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters (e.g., percent change from Baseline). For the primary analysis, OIR was measured when all participants in both treatment arms had two post-Baseline disease assessments. Participants who had an intracranial response of not evaluable or a missing response were treated as non-responders. Confirmation assessments were to be performed no less than 4 weeks after the criteria for response were initially met and may have been performed at the next protocol scheduled assessment.
Time Frame: From the time of the Baseline assessment until disease progression or end of study treatment (average of 18.3 weeks)
Population: V600E Population: all participants with BRAF V600E mutation-positive melanoma who received at least one dose of study treatment
Measure: Number; unit: participants
Groups:
- GSK2118436 150 mg: No Prior Local Therapy: Participants who received no prior local therapy for brain metastasis received GSK2118436 150 mg capsules either one hour before or 2 hours after a meal twice daily until evidence of disease progression, death, or unacceptable adverse events.
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 74 | 65
participants
  CR | 4 | 1
  PR | 26 | 23
Statistical Analysis 1: Comparison: GSK2118436 150 mg: No Prior Local Therapy; Test type: Superiority or Other; p < 0.0001, Exact Test; percentage of participants = 41, 95% CI 2-sided [29.3 to 52.6] — The estimated value represents the percentage of participants with OIR
Statistical Analysis 2: Comparison: GSK2118436 150 mg: Prior Local Therapy; Test type: Superiority or Other; p < 0.0001, Exact Test; percentage of participants = 37, 95% CI 2-sided [25.3 to 49.8] — The estimated value represents the percentage of participants with OIR

2. Secondary Outcome: Number of Participants With V600E Mutation-positive Melanoma With a Best Overall Response (OR) of CR or PR, as Assessed by the Investigator
Description: OR is defined as the number of participants achieving either a CR (the disappearance of all target lesions) or PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]) per modified RECIST, version 1.1. To determine the OR, the extracranial response was combined with the intracranial response. Confirmation assessments were to be performed no less than 4 weeks after the criteria for response were initially met and may have been performed at the next protocol-scheduled assessment. Participants who had an overall response of not evaluable or a missing response were treated as non-responders.
Time Frame: From the time of the Baseline assessment until disease progression or end of study treatment (average of 24 weeks)
Population: V600E Population
Measure: Number; unit: participants
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 74 | 65
participants
  CR | 2 | 0
  PR | 28 | 23

3. Secondary Outcome: Number of Participants With V600K Mutation-positive Melanoma With a Best Overall Response (OR) of CR or PR, as Assessed by the Investigator
Description: as for outcome 2
Time Frame: From the time of the Baseline assessment until disease progression or end of study treatment (average of 17 weeks)
Population: V600K Population: all participants with BRAF V600K mutation-positive melanoma who received at least one dose of study treatment
Measure: Number; unit: participants
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 15 | 18
participants
  CR | 0 | 0
  PR | 0 | 5

4. Secondary Outcome: Number of Participants With V600K Mutation-positive Melanoma With OIR, as Assessed by the Investigator
Description: OIR is defined as the number of participants whose intracranial response was a confirmed complete response (CR) or partial response (PF) assessed by investigators using modified Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters (e.g., percent change from Baseline). For the primary analysis, OIR was measured when all participants in both treatment arms had two post-Baseline disease assessments. Participants who had an intracranial response of not evaluable or a missing response were treated as non-responders. Confirmation assessments were to be performed no less than 4 weeks after the criteria for response were initially met and may have been performed at the next protocol scheduled assessment.
Time Frame: From the time of the Baseline assessment until disease progression or end of study treatment (average of 16 weeks)
Population: V600K Population
Measure: Number; unit: participants
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 15 | 18
participants
  CR | 0 | 0
  PR | 1 | 4

5. Secondary Outcome: Duration of Intracranial Response for the Subset of V600E Mutation-positive Participants
Description: Duration of Intracranial Response is defined as the time from the first documented evidence of intracranial CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]) until the time of the first documented intracranial disease progression (PD) or death due to any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 millimeters (mm).
Time Frame: Time from the first documented evidence of intracranial CR or PR until the time of the first documented intracranial disease progression or death due to any cause (average of 27 weeks)
Population: V600E Population. Only the subset of participants who had a complete or partial intracranial response was included in this analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 30 | 24
weeks | 24.1 [16.1 to 30.3] | 28.1 [24.1 to 44.1]

6. Secondary Outcome: Duration of Intracranial Response for the Subset of V600K Mutation-positive Participants
Description: as for outcome 5
Time Frame: Time from the first documented evidence of intracranial CR or PR until the time of the first documented intracranial disease progression or death due to any cause (average of 31 weeks)
Population: V600K Population. Only the subset of participants who had a complete or partial intracranial response was included in this analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 1 | 4
weeks | 12.4 [NA to NA] — The confidence interval cannot be calculated because too few participants were V600K mutation positive. | NA [16.6 to NA] — The median and the upper limit of the confidence interval cannot be calculated because too few V600K participants had intracranial responses.

7. Secondary Outcome: Duration of Overall Response for the Subset of V600E Mutation-positive Participants
Description: Duration of Overall Response is defined as the time from the first documented evidence of overall CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]) until the time of the first documented disease progression (PD) or death due to any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 millimeters (mm).
Time Frame: Time from the first documented evidence of CR or PR until the time of the first documented disease progression or death due to any cause (average of 28 weeks)
Population: V600E Population. Only the subset of participants who had a complete or partial response was included in this analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 30 | 23
weeks | 27.6 [16.6 to 32.4] | 23.7 [20.0 to 28.1]

8. Secondary Outcome: Duration of Overall Response for the Subset of V600K Mutation-positive Participants
Description: as for outcome 7
Time Frame: Time from the first documented evidence of CR or PR until the time of the first documented disease progression or death due to any cause (average of 31 weeks)
Population: V600K Population. Only the subset of participants who had a complete or partial response was included in this analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 0 | 5
weeks |  | 36.1 [12.3 to NA] — The upper limit of the confidence interval cannot be calculated because too few V600K participants had intracranial responses.

9. Secondary Outcome: Progression-free Survival in V600E Mutation-positive Participants
Description: PFS is defined as the time from the first dose of study medication to the earliest of death or progression (at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 millimeters (mm). If a participant received subsequent anti-cancer therapy prior to the date of documented PD/death, the participant was censored at the last adequate assessment and the visit level response was CR (disappearance of all target lesions), PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters [e.g., percent change from Baseline]), or stable disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Time from the first dose of study medication to the earliest of death or progression (average of 23 weeks)
Population: V600E Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 74 | 65
weeks | 16.1 [15.7 to 23.4] | 16.0 [15.9 to 23.9]

10. Secondary Outcome: Progression-free Survival in V600K Mutation-positive Participants
Description: as for outcome 9
Time Frame: Time from the first dose of study medication to the earliest of death or progression (average of 17 weeks)
Population: V600K Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 15 | 18
weeks | 8.1 [3.1 to 16.1] | 15.6 [7.9 to 17.6]

11. Secondary Outcome: Overall Survival of V600E Mutation-positive Participants
Description: Overall survival (OS) is defined as the time from the first dose of study medication until death due to any cause. OS was censored using the date of last known contact for those participants who were alive at the time of analysis.
Time Frame: Time from the first dose of study medication until death due to any cause (average of 35 weeks)
Population: V600E Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 74 | 65
months | 6.8 [6.1 to 9.2] | 7.6 [6.3 to 10.6]

12. Secondary Outcome: Overall Survival in V600K Mutation-positive Participants
Description: as for outcome 11
Time Frame: Time from the first dose of study medication until death due to any cause (average of 26 weeks)
Population: V600K Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 15 | 18
months | 3.7 [1.6 to 5.2] | 5.0 [3.1 to 11.9]

13. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury.
Time Frame: From Screening until the conclusion of the study (up to 103 weeks)
Population: All Treated Subjects (ATS) Population: all participants who received at least one dose of study treatment
Measure: Number; unit: participants
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 89 | 83
participants
  Any AE | 81 | 79
  Any SAE | 26 | 31

14. Secondary Outcome: Number of Participants With a Worst-case on Therapy Change to Grade 3 and Grade 4, or With Any Grade Increase (AGI), From Baseline Grade for Clinical Chemistry Parameters
Description: Clinical chemistry data were summarized at each scheduled assessment according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE, version 4.0). Grade refers to the severity of the toxicity. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on this general guideline: Grade (G) 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life threatening; Grade 5, death related to toxicity. Blood sample was collected for the assessment of glucose, potassium, magnesium, sodium, phosphorus, potassium. aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), creatinine, total bilirubin, albumin, amylase, cholesterol, creatine kinase, gamma glutamyl transferase (GGT), lipase, blood pH, and triglycerides.
Time Frame: From Screening until the conclusion of the study (up to 103 weeks)
Population: ATS Population. Only those participants with data available for the indicated parameters were analyzed.
Measure: Number; unit: participants
Groups:
- GSK2118436 150 mg: Participants with or without prior local therapy for brain metastasis received GSK2118436 50 mg and 75 mg capsules either one hour before or 2 hours after a meal twice daily.
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 165
participants
  Glucose (hyperglycemia), AGI, n=165 | 71
  Glucose (hyperglycemia), Increase to G 3, n=165 | 8
  Glucose (hyperglycemia), Increase to G 4, n=165 | 1
  Glucose (hypoglycemia), AGI, n=165 | 24
  Glucose (hypoglycemia), Increase to G 3, n=165 | 0
  Glucose (hypoglycemia), Increase to G 4, n=165 | 0
  Magnesium (hypermagnesemia) AGI, n=165 | 2
  Magnesium (hypermagnesemia), Increase to G 3,n=165 | 0
  Magnesium (hypermagnesemia), Increase to G 4,n=165 | 0
  Magnesium (hypomagnesemia), AGI, n=165 | 0
  Magnesium (hypomagnesemia), Increase to G 3, n=165 | 0
  Magnesium (hypomagnesemia), Increase to G 4, n=165 | 0
  Sodium (hypernatremia), AGI, n=165 | 8
  Sodium (hypernatremia), Increase to G 3, n=165 | 0
  Sodium (hypernatremia), Increase to G 4, n=165 | 0
  Sodium (hyponatremia), AGI, n=165 | 21
  Sodium (hyponatremia), Increase to G 3, n=165 | 3
  Sodium (hyponatremia), Increase to G. 4, n=165 | 0
  Phosphorus inorganic, AGI, n=165 | 53
  Phosphorus inorganic, Increase to G 3, n=165 | 13
  Phosphorus inorganic, Increase to G 4, n=165 | 0
  Potassium (hyperkalemia), AGI, n=165 | 8
  Potassium (hyperkalemia), Increase to G 3, n=165 | 0
  Potassium (hyperkalemia), Increase to G 4, n=165 | 0
  Potassium (hypokalemia), AGI, n=165 | 17
  Potassium (hypokalemia), Increase to G 3, n=165 | 4
  Potassium (hypokalemia), Increase to G 4, n=165 | 0
  ALP, AGI, n=165 | 41
  ALP, Increase to G 3, n=165 | 1
  ALP, Increase to G 4, n=165 | 0
  AST, AGI, n=165 | 26
  AST, Increase to G 3, n=165 | 1
  AST, Increase to G 4, n=165 | 0
  ALT, AGI, n=165 | 27
  ALT, Increase to G 3, n=165 | 2
  ALT, Increase to G 4, n=165 | 0
  Creatinine, AGI, n=165 | 10
  Creatinine, Increase to G 3, n=165 | 0
  Creatinine, Increase to G 4, n=165 | 0
  Total bilirubin, AGI, n=163 | 5
  Total bilirubin, Increase to G 3 n=163 | 0
  Total bilirubin, Increase to G 4 n=163 | 0
  Albumin, AGI, n=27 | 9
  Albumin, Increase to G 3, n=27 | 0
  Albumin, Increase to G 4, n=27 | 0
  Amylase, AGI, n=16 | 3
  Amylase, Increase to G 3, n=16 | 1
  Amylase, Increase to G 4, n=16 | 1
  Cholesterol, AGI, n=2 | 1
  Cholesterol, Increase to G 3, n=2 | 0
  Cholesterol, Increase to G 4, n=2 | 0
  Creatine kinase, AGI, n=6 | 1
  Creatine kinase, Increase to G 3, n=6 | 0
  Creatine kinase, Increase to G 4, n=6 | 1
  GGT, AGI, n=22 | 13
  GGT, Increase to G 3, n=22 | 4
  GGT, Increase to G 4, n=22 | 0
  Lipase, AGI, n=19 | 10
  Lipase, Increase to G 3, n=19 | 4
  Lipase, Increase to G 4, n=19 | 2
  Blood pH, AGI, n=1 | 0
  Blood pH, Increase to G 3, n=1 | 0
  Blood pH, Increase to G 4, n=1 | 0
  Triglycerides, AGI, n=5 | 3
  Triglycerides, Increase to G 3, n=5 | 0
  Triglycerides, Increase to G 4, n=5 | 0

15. Secondary Outcome: Number of Participants With the Indicated Hepatobiliary Laboratory Abnormalities
Description: Blood samples were collected for the assessment of hepatobiliary parameters. ALT=alanine aminotranserase; AST=aspartate aminotransferase; ALP=alkaline phosphatase; BIL=total bilirubin; INR=international normalized ratio; ULN=upper limit of normal. Hepato-cellular injury is defined as (ALT/ULN)/(ALP/ULN) >=5.
Time Frame: From Screening until the conclusion of the study (up to 103 weeks)
Population: ATS Population
Measure: Number; unit: participants
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 89 | 83
participants
  Possible HYs Law, >3x ULN ALT, >=2x ULN BIL | 0 | 0
  Possible HYs Law, >3x ULN ALT, >1.5x ULN INR | 0 | 0
  Hepato-cellular injury | 2 | 1
  Bilirubin elevations, >=2x ULN BIL | 0 | 1
  Bilirubin elevations, >=2x ULN BIL and <2x ULN BIL | 0 | 1
  ALT or AST elevations, >3x ULN ALT or AST | 2 | 4
  ALT or AST elevations, >5x ULN ALT or AST | 1 | 1
  ALT or AST elevations, >8x ULN ALT or AST | 1 | 1
  ALT or AST elevations, >20x ULN ALT or AST | 0 | 0
  ALT elevations, >3x ULN ALT | 2 | 4
  ALT elevations, >5x ULN ALT | 1 | 1
  ALT elevations, >8x ULN ALT | 1 | 1
  ALT elevations, >20x ULN ALT | 0 | 0
  ALT elevations, >3x ULN ALT, <=3x ULN ALT Baseline | 2 | 4
  ALP elevations, >=3x ULN ALP | 5 | 2
  ALP elevations, >=3x ULN ALP and <3x ULN ALP | 4 | 2

16. Secondary Outcome: Number of Participants With a Worst-case on Therapy Change to Grade 3 and Grade 4, or With Any Grade Increase (AGI), From Baseline Grade for Hematology Parameters
Description: Hematology data were summarized at each scheduled assessment according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE, version 4.0). Grade refers to the severity of the toxicity. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on this general guideline: Grade 1, mild; Grade 2, moderate; Grade 3, severe, Grade 4, life threatening, Grade 5, death related to toxicity. Blood sample was collected for the assessment of hemoglobin, white blood cells, and platelet count.
Time Frame: From Screening until the conclusion of the study (up to 103 weeks)
Population: ATS Population. Only those participants with data available for the indicated parameters were analyzed.
Measure: Number; unit: participants
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 84 | 81
participants
  Hemoglobin (anemia), AGI | 25 | 81
  Hemoglobin (anemia), Increase to Grade 3 | 2 | 3
  Hemoglobin (anemia), Increase to Grade 4 | 0 | 0
  Hemoglobin (increased), AGI | 1 | 0
  Hemoglobin (increased), Increase to Grade 3 | 0 | 0
  Hemoglobin (increased), Increase to Grade 4 | 0 | 0
  Lymphocyte count increased, AGI | 0 | 0
  Lymphocyte count increased, Increase to Grade 3 | 0 | 0
  Lymphocyte count increased, Increase to Grade 4 | 0 | 0
  Lymphocyte count decreased, AGI | 18 | 81
  Lymphocyte count decreased, Increase Grade 3 | 4 | 6
  Lymphocyte count decreased, Increase Grade 4 | 1 | 0
  Total neutrophils, AGI, | 6 | 11
  Total neutrophils, Increase to Grade 3 | 0 | 0
  Total neutrophils, Increase to Grade 4 | 2 | 2
  Platelet count, AGI | 7 | 9
  Platelet count, Increase to Grade 3 | 2 | 1
  Platelet count, Increase to Grade 4 | 1 | 0
  White blood cell count, AGI | 9 | 16
  White blood cell count, Increase to Grade 3 | 0 | 0
  White blood cell count, Increase to Grade 4 | 1 | 1

17. Secondary Outcome: Mean Blood Pressure at Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, and 36
Description: Systolic and diastolic blood pressure were measured for all treated participants.
Time Frame: Baseline; Weeks 4, 8, 12, 16, 20, 24, 28, 32, and 36
Population: ATS Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 89 | 83
millimeters of mercury (mmHg)
  Diastolic BP, Baseline, n=89,83 | 77.7 (8.78) | 77.1 (9.73)
  Diastolic BP, Week 4, n=81, 78 | 74.0 (10.12) | 74.6 (10.88)
  Diastolic BP, Week 8, n=70, 73 | 74.6 (9.14) | 72.7 (9.54)
  Diastolic BP, Week 12, n=68, 62 | 75.2 (7.70) | 74.3 (11.64)
  Diastolic BP, Week 16, n=52, 52 | 73.2 (10.01) | 71.4 (9.40)
  Diastolic BP, Week 20, n=29, 34 | 73.6 (9.98) | 71.7 (9.67)
  Diastolic BP, Week 24, n=22, 25 | 74.7 (7.87) | 72.7 (9.99)
  Diastolic BP, Week 28, n=15, 17 | 73.9 (6.98) | 76.5 (8.37)
  Diastolic BP, Week 32, n=9, 7 | 73.1 (9.47) | 73.6 (9.64)
  Diastolic BP, Week 36, n=2, 1 | 75.5 (7.78) | 93.0 (NA) — Standard deviation could not be calculated because only one participant was analyzed in this treatment group at this time point.
  Systolic BP, Baseline, n=89, 83 | 126.6 (16.73) | 123.9 (14.17)
  Systolic BP, Week 4, n=81, 78 | 122.2 (13.68) | 121.9 (15.37)
  Systolic BP, Week 8, n=70, 73 | 123.0 (12.71) | 117.3 (14.53)
  Systolic BP, Week 12, 68, 62 | 123.6 (14.74) | 120.1 (14.21)
  Systolic BP, Week 16, n=52, 52 | 124.7 (17.70) | 119.9 (11.67)
  Systolic BP, Week 20, n=29, 34 | 123.7 (16.02) | 118.9 (13.51)
  Systolic BP, Week 24, n=22, 25 | 126.3 (17.80) | 120.9 (16.63)
  Systolic BP, Week 28, n=15, 17 | 122.2 (17.03) | 120.8 (14.32)
  Systolic BP, Week 32, n=9, 7 | 122.8 (14.84) | 117.7 (10.01)
  Systolic BP, Week 36, n=2, 1 | 119.5 (13.44) | 128.0 (NA) — Standard deviation could not be calculated because only one participant was analyzed in this treatment group at this time point.

18. Secondary Outcome: Number of Participants With a Worst-case On-therapy Increase From Baseline in Bazett's QTc Reading in the 12-lead Electrocardiogram (ECG)
Description: An increase in the QTc interval corrected using Bazett's formula (Bazett's QTc) was recorded for all treated participants. Grade 1 (450-480 milliseconds [msec]), Grade 2 (481-500 msec), Grade 3/4 (>=501 msec). An increase is defined as an increase in CTCAE grade relative to Baseline grade.
Time Frame: Baseline; Weeks 4, 12, 20, 28, 40, 52, and 64
Population: ATS Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 75 | 74
participants
  Increase from Baseline to any grade | 11 | 17
  Increase from Baseline to Grade 2 | 1 | 2
  Increase from Baseline to Grade 3/4 | 0 | 0

19. Secondary Outcome: Number of Participants With Abnormal Echocardiograms (ECHO) at Weeks 4 and 12
Description: Echocardiograms (ECHO) were measured for all treated participants. An echocardiogram test gives information about the structure and function of the heart. LLN=lower limit of normal (determined by the institution).
Time Frame: Weeks (W) 4 and 12
Population: ATS Population
Measure: Number; unit: participants
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 89 | 83
participants
  W 4, Left ventricle (LV) ejection fraction < LLN | 1 | 0
  W 4, LV ejection fraction < normal | 0 | 0
  W 12, LV ejection fraction < LLN | 0 | 0
  W 12, LV ejection fraction < normal | 1 | 0

20. Secondary Outcome: Median Concentrations of GSK2118436 and Its Metabolites Including GSK2285403, GSK2298683, and GSK2167542
Description: Summary statistics were calculated for each time point by cohort. The population pharmacokinetics were determined using a non-linear mixed effects modeling approach after pooling the data with other studies. These results are reported separately.
Time Frame: Week 4 (pre-dose and 1-3 hours post-dose) and Weeks 8, 16, 24, and 32 (either pre-dose in the morning or in the afternoon at 4-8 hours post-dose)
Population: PK Population: participants in the ATS population for whom a PK sample was obtained and analyzed. Only those participants whose samples were available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: nanograms per milliliter (ng/mL)
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 75 | 77
nanograms per milliliter (ng/mL)
  GSK2118436, Week 4, predose, n=55, 58 | 31.6 [7 to 2995] | 50.2 [0 to 4293]
  GSK2118436, Week 4, 1-3 hours (hrs), n=63, 70 | 992.1 [5 to 4870] | 810.7 [4 to 4995]
  GSK2118436, Week 8, predose, n=36, 36 | 27.2 [8 to 1148] | 37.5 [3 to 944]
  GSK2118436, Week 8, 4-8 hrs, n=19, 25 | 274.7 [28 to 1062] | 294.5 [15 to 2011]
  GSK2118436, Week 16, predose, n=26, 23 | 27.8 [6 to 3390] | 30.7 [3 to 203]
  GSK2118436, Week 16, 4-8 hrs, n=11, 18 | 341.5 [33 to 1141] | 295.8 [55 to 1808]
  GSK2118436, Week 24, predose, n=14, 10 | 60.7 [1 to 597] | 53.8 [14 to 211]
  GSK2118436, Week 24, 4-8 hrs, n=5, 12 | 371.2 [0 to 1072] | 226.1 [30 to 974]
  GSK2118436, Week 32, predose, n=11, 7 | 38.6 [7 to 777126] | 28.4 [2 to 87]
  GSK2118436, Week 32, 4-8 hrs, n=2, 8 | 227.6 [90 to 365] | 335.7 [94 to 1939]
  GSK2285403, Week 4, predose, n=55, 58 | 62.7 [9 to 1495] | 80.5 [0 to 2931]
  GSK2285403, Week 4, 1-3 hrs, n=63, 70 | 688.9 [15 to 2499] | 593.2 [8 to 2812]
  GSK2285403, Week 8, predose, n=36, 36 | 46.5 [10 to 1743] | 74.4 [6 to 553]
  GSK2285403, Week 8, 4-8 hrs, n=19, 25 | 335.5 [55 to 1114] | 310.5 [12 to 3160]
  GSK2285403, Week 16, predose, n=26, 23 | 45.1 [10 to 824] | 54.4 [5 to 354]
  GSK2285403, Week 16, 4-8 hrs, n=11, 18 | 434.1 [44 to 976] | 456.9 [148 to 1053]
  GSK2285403, Week 24, predose, n=14, 10 | 97.3 [6 to 386] | 103.3 [14 to 325]
  GSK2285403, Week 24, 4-8 hrs, n=5, 12 | 617.1 [0 to 1057] | 357.7 [79 to 959]
  GSK2285403, Week 32, predose, n=11, 7 | 63.1 [8 to 934] | 46.6 [4 to 88]
  GSK2285403, Week 32, 4-8 hrs, n=2, 8 | 375.3 [118 to 633] | 377.5 [117 to 1519]
  GSK2298683, Week 4, predose, n=55, 58 | 3215.8 [1225 to 14064] | 3877.4 [43 to 13435]
  GSK2298683, Week 4, 1-3 hrs, n=63, 70 | 4272.5 [747 to 18161] | 4500.3 [275 to 18196]
  GSK2298683, Week 8, predose, n=36, 36 | 3152.0 [1564 to 10402] | 3250.0 [667 to 12747]
  GSK2298683, Week 8, 4-8 hrs, n=19, 25 | 4692.1 [2133 to 11320] | 5447.5 [2015 to 15009]
  GSK2298683, Week 16, predose, n=26, 23 | 3070.0 [1143 to 11414] | 3561.2 [922 to 10204]
  GSK2298683, Week 16, 4-8 hrs, n=11, 18 | 4865.5 [2670 to 11821] | 6595.7 [1630 to 11380]
  GSK2298683, Week 24, predose, n=14, 10 | 3026.8 [1532 to 14762] | 4199.7 [2040 to 7504]
  GSK2298683, Week 24, 4-8 hrs, n=5, 12 | 3825.9 [320 to 13056] | 5659.9 [3225 to 11009]
  GSK2298683, Week 32, predose, n=11, 7 | 2386.6 [1421 to 6528] | 2451.7 [1253 to 5026]
  GSK2298683, Week 32, 4-8 hrs, n=2, 8 | 11225.8 [5323 to 17129] | 6547.4 [4578 to 8786]
  GSK2167542, Week 4, predose, n=55, 58 | 317.9 [50 to 1338] | 323.0 [3 to 2690]
  GSK2167542, Week 4, 1-3 hrs, n=63, 70 | 351.6 [62 to 1505] | 332.1 [46 to 1619]
  GSK2167542, Week 8, predose, n=36, 36 | 324.1 [86 to 964] | 298.6 [56 to 1272]
  GSK2167542, Week 8, 4-8 hrs, n=19, 25 | 305.4 [91 to 899] | 320.5 [78 to 960]
  GSK2167542, Week 16, predose, n=26, 23 | 285.5 [93 to 1095] | 310.8 [35 to 1200]
  GSK2167542, Week 16, 4-8 hrs, n=11, 18 | 291.1 [69 to 769] | 320.5 [81 to 652]
  GSK2167542, Week 24, predose, n=14, 10 | 304.0 [94 to 875] | 334.0 [63 to 795]
  GSK2167542, Week 24, 4-8 hrs, n=5, 12 | 190.7 [19 to 401] | 287.9 [106 to 599]
  GSK2167542, Week 32, predose, n=11, 2 | 361.2 [113 to 960] | 316.3 [69 to 690]
  GSK2167542, Week 32, 4-8 hrs, n=2, 8 | 227.8 [225 to 231] | 273.9 [231 to 1021]

21. Secondary Outcome: Composite of Pharmacokinetic Parameters of GSK2118436 in a Subset of Participants Receiving Dexamethasone
Description: This outcome measure could not be analyzed because too few participants participated in the dexamethasone study.
Time Frame: Day 15
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Number of Response Genetics Incorporated (RGI) Investigational Use Only (IUO) Assay Mutation Positive Participants and THxID BRAF Assay Mutation Positive Participants With the Indicated Best Intracranial Response
Description: The BRAF screening assay determines the specific BRAF mutational status (V600 E and K) in participants with metastatic melanoma who may benefit from treatment with GSK2118436. Per RECIST, version 1.1, CR is defined as the disappearance of all lesions. PR is defined as a >=30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline (BL) sum of the diameters (e.g., percent change from BL). Stable disease is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD is defined as a >=20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir [smallest sum of diameters recorded since treatment start]). In addition, the sum must have an absolute increase from nadir of 5 millimeters. Not evaluable: cannot be classified by a preceding definition.
Time Frame: Screening
Population: V600EK and THIDEK Population: all enrolled participants who were V600E or V600K mutation positive by the RGI IUO assay
Measure: Number; unit: participants
Groups:
- RGI IUO Mutation Positive Participants: Melanoma participants determined to be positive for the BRAF V600E and V600K mutations as determined by the RGI assay. The RGI assay is a BRAF mutation test developed by Response Genetics Incorporated, and was used to determine eligibility. It employs the allele-specific polymerase chain reaction (ASPCR) methodology, and was offered as an Investigational Use Only assay (only for pre-market investigational purposes).
- ThxID BRAF Mutation Positive Participants: Melanoma participants determined to be positive for the BRAF V600E and V600K mutations as determined by the ThxID assay. The RGI test was further validated by BioMerieux (BMX THxID assay) for regulatory approval. The THxID IUO assay was used to retrospectively confirm the RGI test results.
Arm/Group | RGI IUO Mutation Positive Participants | ThxID BRAF Mutation Positive Participants
Number analyzed (Participants) | 172 | 155
participants
  Complete response | 2 | 2
  Partial response | 52 | 49
  Stable disease | 78 | 69
  Progressive disease | 26 | 23
  Not evaluable | 14 | 12

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the time the first dose of study treatment was administered until 30 days following discontinuation of study treatment (up to 103 weeks).
Description: SAEs and non-serious AEs were collected in the All Treated Subjects (ATS) Population, comprised of all participants who received at least one dose of study medication.
Arm/Group | GSK2118436 150 mg: No Prior Local Therapy | GSK2118436 150 mg: Prior Local Therapy
Serious Adverse Events (participants affected / at risk) | 26/89 | 31/83
Other Adverse Events (participants affected / at risk) | 79/89 | 74/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2118436 150 mg: No Prior Local Therapy (N=89) | GSK2118436 150 mg: Prior Local Therapy (N=83)
Pyrexia (Gastrointestinal disorders) | 4 | 9
Haemorrhage intracranial (Nervous system disorders) | 2 | 3
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7
Headache (Nervous system disorders) | 2 | 2
Chills (General disorders) | 1 | 2
Hypotension (Vascular disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 2 | 0
Ejection fraction decreased (Investigations) | 3 | 0
Fatigue (General disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Viral pericarditis (Infections and infestations) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 1
Intracranial tumour haemorrhage (Nervous system disorders) | 1 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2118436 150 mg: No Prior Local Therapy (N=89) | GSK2118436 150 mg: Prior Local Therapy (N=83)
Headache (Nervous system disorders) | 24 | 20
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 24 | 20
Nausea (Gastrointestinal disorders) | 16 | 26
Pyrexia (General disorders) | 23 | 15
Fatigue (General disorders) | 18 | 25
Vomiting (Gastrointestinal disorders) | 18 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 13
Rash (Skin and subcutaneous tissue disorders) | 16 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 15 | 10
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 | 8
Diarrhoea (Gastrointestinal disorders) | 7 | 15
Decreased appetite (Metabolism and nutrition disorders) | 8 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 8
Chills (General disorders) | 9 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 5
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 7
Constipation (Gastrointestinal disorders) | 3 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 4
Insomnia (Psychiatric disorders) | 6 | 6
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 4
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4
Anaemia (Blood and lymphatic system disorders) | 6 | 4
Alanine aminotransferase increased (Investigations) | 6 | 4
Oedema peripheral (General disorders) | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 2
Asthenia (General disorders) | 2 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 | 3
Dizziness (Nervous system disorders) | 5 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 3
Lymphopenia (Blood and lymphatic system disorders) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Confusional state (Psychiatric disorders) | 0 | 7
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Nasopharyngitis (Infections and infestations) | 5 | 2
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 6
Depression (Psychiatric disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.